CLINICAL TRIAL: NCT07201207
Title: Single-center, Randomized, Controlled, Double Blinded, 24-month Trial to Compare Robotic-assisted (MAKO) and Manual Total Knee Arthroplasty for Primary Osteoarthritis With 10 Year Follow-up for Complications
Brief Title: Robotic-assisted (MAKO) Versus Manual Total Knee Arthroplasty for Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satakunta Central Hospital (Other)
Responsible Party: Principal Investigator, Juha Kukkonen, Docent, MD, Satakunta Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VARHA/28584/13.02.02/2024
Record Dates: First submitted 2025-08-28; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Knee
Keywords: arthroplasty; robotic-assisted arthroplasty; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic-assisted total knee arthroplasty (Experimental): The intervention group will undergo MAKO assisted RATKA. The patients will have individualized alignment. Knee balance is achieved with bony cuts and implant positioning, to avoid soft tissue releases. A preoperative planning based on computed tomography (CT) scans is made and intraoperatively computer assisted gap balancing is performed based on the plan and patient's soft tissue envelope and native joint line. The precise pre-operative planning, balancing and alignment method has been described by Calliess T el al.
  Interventions: Device: Robotic-assisted total knee arthroplasty
- Manual total knee arthroplasty (Active Comparator): The control group will undergo manual jig-guided TKA, with bony cuts made to achieve neutral mechanical axis, and if necessary, knee balancing will be performed by soft tissue releases. Weight bearing semi-flexion radiographs and long leg radiographs are used for preoperative planning. Intramedullary guiding rod is used in femur to align the cuts in 6 to 7 degrees of valgus. Femoral component rotation is fixed to trans-epicondylar line. Tibia cuts are aligned with either intra- or extramedullary guiding rod according to the preference of the surgeon. Tibia component rotation is fixed to medial one-third of tibial tubercle. After bony cuts, knee balancing is performed with soft-tissue and ligament releases if necessary.
  Interventions: Procedure: Manual total knee arthroplasty

INTERVENTIONS:
Device: Robotic-assisted total knee arthroplasty — In robotic-assisted total knee arthroplasty, the procedure is performed with the guidance of the robot according to CT-based plan.
  Arms: Robotic-assisted total knee arthroplasty
Procedure: Manual total knee arthroplasty — In manual total knee arthroplasty, the procedure is performed with jig guides according to whole leg weight bearing x-ray planning.
  Other Names: Traditional total knee arthroplasty; Jig-guided total knee arthroplasty
  Arms: Manual total knee arthroplasty

SUMMARY:
Background: Total knee arthroplasty is a golden standard procedure for end-stage knee osteoarthritis. However, up to 20% of the patients are not satisfied with the outcome. Recently, robotic-assisted TKAs have been developed to offer individual alignment and to achieve accuracy in positioning with more subtle soft-tissue handling, thus possibly leading into better outcome.

Hypothesis: The investigators hypnotize that, robotic-assisted TKA is superior to manual TKA for end-stage osteoarthritis in respect to functional outcome, short-term rehabilitation and cost-efficiency.

Trial desing: The investigators will conduct a single-center, randomized, controlled, double blinded superiority trial of 24-months to compare robotic-assisted and manual total knee arthroplasty in respect to functional outcome, implant positioning, short-term rehabilitation and cost-efficiency with up to 10 years follow-up for complications.

The principle outcome measure will be patient reported outcome measure (PROM) Oxford knee score (OKS) points (0-48 points) at two years after surgery. Minimal clinically important difference will be considered as 5 points. Other PROMS, patient satisfaction, short-term rehabilitation, implant positioning, knee range of motion, length of sick leave and cost efficiency will also be reported. Patients will be followed up to 10 years for complications (infection, manipulation and revisions).

This study will be conducted in Central Hospital of Satakunta (Satasairaala), Finland. The investigators will recruit 170 adult patients (aged 50-80), with end-stage (Kellgren-Lawrence grade IV) primary osteoarhritis. Patients will be randomly assingned to either robotic-assisted or manual TKA. Patients will be blinded by the intervention method used. Personnel and investigators assessing the patients and interpreting the data will also be blinded to the surgical method.

ELIGIBILITY:
Inclusion criteria

* Age over 50 and below 80 years
* End-stage Kellgren-Lawrence grade IV KOA
* Failed conservative treatment

Exclusion criteria

* Post-traumatic knee osteoarthritis
* Rheumatoid arthritis
* Previous knee infections
* Previous knee surgery (other than diagnostic arthroscopy or meniscectomy)
* Knee range of motion within 15 to 100 degrees
* Mechanical axis over 15 degrees of varus or over 10 degrees of valgus
* Body mass index over 40 kg/m2
* Significant patellofemoral osteoarthritis (Kellgren-Lawrence grade III or IV)
* Diabetes treated with insulin
* Malignancy with ongoing treatment
* Systemic glukocorticosteroid or antimetabolite medication during the last 5 years
* Conditions that do not allow general anesthesia
* Patients' denial for operative treatment and/or participation in the trial

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2037-09 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee score OKS at 24 months | 24 month
  Patient reported outcome measure, knee function questionnaire Oxford Knee Score (OKS) at 24 month. Scale from 0 (=worst) to 48 (=excellent) points Minimal clinically important difference considered as 5 points.

SECONDARY OUTCOMES:
Oxford Knee Score at 3 and 12 months | 3 and 12 months visits
  Patient reported outcome measure, knee function questionnaire Oxford Knee Score (OKS) at 3 and 12 months. Scale from 0 (=worst) to 48 (=excellent) points. Minimal clinically important difference considered as 5 points.
Knee injury and Osteoarthritis Outcome Score (KOOS) at 3, 12 and 24 months | 3, 12 and 24 months
  Patient reported outcome measure, knee function questionnaire KOOS points at 3, 12 and 24 months after the operation. Scale from 0 (=worst) to 100 (=excellent).
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) at 3, 12 and 24 months. | 3, 12 and 24 months
  Patient reported outcome measure, knee function questionnaire WOMAC score at 3, 12 and 24 months after the operation. Scale from 0 (= excellent) to 96 (= worst) points.
Patient satisfaction inquiry at 3, 12 and 24 months | 3, 12 and 24 months
  Patient satisfaction question asked at 3, 12 and 24 months after the operation: If you could choose again, would you still go for the sugery? 0= no 1 = probably not 2= I don't know 4 = probably yes 5 = yes.
Working ability, lenght of the sick leave | up to 24 months
  Length of the sick leave after the surgery, measured as days. Asked from the patient and checked from the patient files.
Working ability, part-time vs full-time | Asked at 3 month, 12 months and 24 months after the surgery
  Asked from the patient at the 3, 12 and 24 months follow-ups visits. Has the operation changed your ability to work full-time or part-time? Options: a) yes my work changed from full-time to part-time after surgery b) no my work is as much full-time or part-time as it was before the surgey c) yes my work changed from full-time to part-time after surgery d) my work as part-time or full-time has changed from other reasons not related to the knee.
Working ability, physical demands of the job | Asked at 3 month, 12 months and 24 months after the surgery
  Asked from the patient at the 3, 12 and 24 months follow-ups visits. Has the physical demands of your job changed after the operation because of the knee? Options: a) yes the physical demands of my job is now lower than it was before the surgery b) no my work is as physically demanding as it was before the surgery c) yes the physical demands of my job is now higher than it was before the surgery d) the physical demands of my job has changed from other reasons not related to the knee.
Life quality questionnaire 15 dimensions (15D) at 3, 12 and 24 months | 3, 12 and 24 months
  Life quality questionnaire 15 dimensions at 3 follow up visits. Scale from 15 (=exellent) to 75 (=worst) points.
Pain at rest and during walking on visual analoque scale (VAS) | First day after the operation and at 3, 12 and 24 months
  pain at rest and during walking on visual analoque scale (VAS) from 0 (=no pain) to 10 (=extreme pain)
Opioid usage | Up to two weeks
  Opioid usage mg/day
Blood loss | First day after the operation
  Blood loss evaluated by the by measuring pre- and post-operative (first day after surgery) hemoglobin g/L. Difference between the pre-operative and post-operative Hemoglobin (g/L) values.
Lenght of the hospital stay | Up to 1 week
  Length of hospital stay measured in days.
Operation time | Day of the surgery
  Time of the operation in hours and minutes checked form patient files.
Post-operative CRP | First day after the operation
  post-op CRP as a indirect soft-tissue damage measure
Knee swelling | First day after the operation
  Knee swelling, knee diameter measured above the patella and compared to the unaffected size, the diameter difference in centimeters between the legs. Indirect soft-tissue damage measures
Range of knee motion (ROM) | First day after the operation and at 3, 12 and 24 months visits
  Range of knee motion measured with goniometry as degrees at the ward on first post-operative day and ant the 3, 12 and 24 months visits.
Radiological outcome measures, alingment | Weight bearing whole leg x-rays taken 3 months post-operatively.
  Knee alignment measured from post-operative weight bearing whole leg x-rays as degrees. Measured as the degrees between femoral mechanical axis line and tibial mechanical axis line.
Radiological outcome measures, posterior condylar offset | post-operative knee x-rays taken within 1 week after the operation
  Post-op knee x-ray taken at the first post-operative day; posterior condylar offset, measured as maximal thickness of the posterior condyle projecting posteriorly to a straight line drawn as the extension of the posterior femoral shaft cortex, measured in millimeters
Radiological outcome measures, Insall-salvati ratio | post-operative knee x-rays taken within 1 week after the operation
  Measured from post-operative knee x-rays. Insall-salvati ratio: the length of the patellar tendon in millimeters divided by the length of the patella in millimeters.
Radiological outcome measures, Overhanging | post-operative knee x-rays taken within 1 week after the operation
  Measured from post-operative knee x-rays. Overhanging of the tibial or femoral component from medial lateral, posterior or anterior side measured as millimeters. The length between the bony edge to the edge of the component.
Radiological outcome measures, Notching | post-operative knee x-rays taken within 1 week after the operation
  Measured from post-operative knee x-rays. Notching of the anterior femoral cortex. The lenght in millimeters between the anterior femoral cortex and the anterior edge femoral component in sagittal x-ray.
Complications, revisons | 3, 12 and 24 months and five and ten years
  Revisions meaning re-operation of the knee due any reason. Checked from the patient files at 3, 12 and 24 months and five and ten years after surgery. Measured as number of revisions
Complications, infections | 3, 12 and 24 months and five and ten years after surgery
  Infections that recuire antibiotics or revision surgery. Checked from the patient files at 3, 12 and 24 months and five and ten years after surgery. Measured as number of infections
Complications, knee manipulation under anestesia due stiff knee | 3, 12 and 24 months and five and ten years after surgery.
  Need for knee manipulations under anesthesia due stiff knee. Measured as number of manipulations. Checked form the patient files at 3, 12 and 24 months and five and ten years after surgery
Complications, re-admission | up to 24 months
  Unplanned post-operative re-admissions due to the knee operation. Measured as days at the ward.
Complications, unplannet emergency unit visits | up to 24 months
  Unplanned post-operative visits to the hospital emergency unit due to the knee operation, number of visits
Costs | up to 24 months
  Total cost of the treatment, measured as amount of money.

CONTACTS AND LOCATIONS:
Overall Officials: Silja Voutilainen, MD, PhD, Study Chair — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No